CLINICAL TRIAL: NCT05944874
Title: Effect of Non-invasive Neurostimulation on Variability of Heart Rate During the Six-minute Walk Test of Patients With Heart Failure: a Double-blinded Clinical Trial
Brief Title: Effect of Non-invasive Neurostimulation on Variability OF HEART RATE IN PATIENTS WITH HEART FAILURE.
Acronym: HD-tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, José Heriston de Morais Lima, teacher, Federal University of Paraíba
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 64878922.2.0000.5188
Record Dates: First submitted 2023-06-14; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
Keywords: Heart failure; transcranial direct current stimulation; six minute walk test
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This study is a clinical trial, and may also be called a "before and after" study, in which all subjects receive the same treatment and their condition is checked before beginning and after various moments of treatment
Who Masked: Participant, Care Provider, Investigator
Masking Description: HD-TDCS applicator, six-minute walk test evaluator, and patient are blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HD- TDCS (inhibition) (Experimental): Patients will perform a session (inhibition) of HD-TDCS of twenty minutes with intensity of 3 milliamps in the left temporal cortex. Before and after each session, patients will perform the six-minute walk test. Heart rate variability (HRV) will be evaluated throughout the protocol through Holter (3-channel). At the end, the perception of exertion and the level of dyspnea of the patient, distance covered and blood pressure will be evaluated.
  Interventions: Device: high definition transcranial direct current stimulation
- HD- TDCS (stimulation) (Experimental): Patients will perform a session (stimulation) of HD-TDCS of twenty minutes with intensity of 3 milliamps in the left temporal cortex. Before and after each session, patients will perform the six-minute walk test. Heart rate variability (HRV) will be evaluated throughout the protocol through Holter (3-channel). At the end, the perception of exertion and the level of dyspnea of the patient, distance covered and blood pressure will be evaluated.
  Interventions: Device: high definition transcranial direct current stimulation
- HD- TDCS (shan) (Experimental): Patients will perform a twenty-minute session (SHAN) of HD-TDCS with an intensity of 3 milliamps in the left temporal cortex. Before and after each session, patients will perform the six-minute walk test. Heart rate variability (HRV) will be evaluated throughout the protocol through Holter (3-channel). At the end, the perception of exertion and the level of dyspnea of the patient, distance covered and blood pressure will be evaluated.
  Interventions: Device: high definition transcranial direct current stimulation

INTERVENTIONS:
Device: high definition transcranial direct current stimulation — Transcranial direct current stimulation, in recent decades, has been identified as a non-invasive tool for transiently modulating human brain activity. The technique consists of the application of a low-intensity continuous electric current, through electrodes applied to the scalp, acting in a regulatory way on the frequency of triggered action potentials, however, without interacting directly with the neurons.
  Other Names: HD-tDCS

SUMMARY:
This study is a clinical trial, and may also be referred to as a "before and after" study, in which all subjects receive the same treatment and their condition is checked before initiation and after various times of treatment. This study will be carried out at the Laboratory of Physiotherapy in Cardiorespiratory Research, located in the building of the postgraduate course in physiotherapy at the Health Sciences Center (CCS) of the Federal University of Parahyba (UFPB), from May 2023 to May 2020. 2024. After screening, patients will undergo assessment and anthropometric measurements. Subsequently, interventions will be carried out

DETAILED DESCRIPTION:
The patients will perform three sessions of HD-TDCS (stimulation, inhibition and Shan) of twenty minutes with an intensity of three milliamps in the left temporal cortex. Before and after each session, patients will perform the six-minute walk test. Heart rate variability (HRV) will be evaluated throughout the protocol through Holter (3-channel). At the end, the perception of exertion and the level of dyspnea of the patient, distance covered and blood pressure will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of heart failure;
* over eighteen years old;
* classified in functional class II and III of the New York Heart Association.

Exclusion Criteria:

* Patients with neurological or pulmonary diseases;
* Patients with cognitive alterations that make it impossible to execute commands;
* with physical limitations that prevent the performance of the exercise protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Travelled distance | day one
  To analyze the distance walked by these patients after the six-minute walk test after the application of HD-Tdcs
heart rate variability | day one
  To evaluate the effects of HD-TDCS on the left temporal lobe - T3 on heart rate variability during the six-minute walk test in patients with heart failure

CONTACTS AND LOCATIONS:
Overall Officials: José Sr Heriston, Principal Investigator — Federal University of Paraiba
Locations (1):
- University Hospital Lauro Wanderley, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No